CLINICAL TRIAL: NCT00507689
Title: A Phase 2, Open-Label Randomized Study to Evaluate the Efficacy and Safety of the Combination Product, Emtricitabine/Tenofovir Disoproxil Fumarate in the Presence or Absence of Hepatitis B Immunoglobulin (HBIg) in Preventing Recurrence of Chronic Hepatitis B (CHB) Post-Orthotopic Liver Transplant (OLT)
Brief Title: Truvada Versus Truvada Plus Hepatitis B Immunoglobulin (HBIg) in Prevention of Chronic Hepatitis B Recurrence Post Liver Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GS-US-203-0107
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Results first posted 2013-09-19 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Hepatitis B
Keywords: Truvada; HBIg; Chronic Hepatitis B Recurrence; Post Orthotopic Liver Transplant
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; hepatitis B hyperimmune globulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FTC/TDF+HBIg (Experimental): Participants received FTC/TDF+HBIg for up to 24 weeks in the pre-randomization period; those who completed 24 weeks of treatment were then randomized to receive FTC/TDF+HBIg in the randomized period.
  Interventions: Drug: FTC/TDF; Drug: Hepatitis B Immunoglobulin (HBIg)
- FTC/TDF (Experimental): Participants received FTC/TDF+HBIg for up to 24 weeks in the pre-randomization period; those who completed 24 weeks of treatment were then randomized to receive FTC/TDF in the randomized period.
  Interventions: Drug: FTC/TDF

INTERVENTIONS:
Drug: FTC/TDF — Emtricitabine (FTC) 200 mg/tenofovir disoproxil fumarate (TDF) 300 mg was administered as a fixed-dose combination tablet orally once daily.
  Other Names: Truvada
Drug: Hepatitis B Immunoglobulin (HBIg) — HBIg was administered either intravenously or by intramuscular injection at a dose and frequency as prescribed by the investigative site protocol.
  Arms: FTC/TDF+HBIg

SUMMARY:
The objective of this 96-week study was to evaluate the safety and antiviral efficacy of emtricitabine/tenofovir disoproxil fumarate (FTC/TDF, coformulated; Truvada®) with or without hepatitis B immunoglobulin (HBIg) in preventing the recurrence of chronic hepatitis B following liver transplantation, in participants who were chronically infected with hepatitis B prior to transplantation.

Prior to enrollment, participants were required to have received at least 12 weeks of HBIg therapy following liver transplantation. Enrolled participants then received FTC/TDF plus HBIg for an initial 24-week pre-randomization treatment period. Participants who completed the pre-randomization period and who achieved sustained viral suppression were randomized to continue treatment with FTC/TDF with or without HBIg for an additional 72 weeks (randomized period). The antiviral efficacy of treatment was assessed by measuring hepatitis B virus levels in the blood (HBV DNA). Safety and tolerability was monitored by assessing adverse events and various laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18-75 years of age) with either hepatitis e antigen (HBeAg) positive or HBeAg negative chronic HBV prior to transplant
* Willing and able to provide written informed consent
* Subjects with detectable antibody to hepatitis B surface antigen performed by a local laboratory result within 30 days of screening
* Subjects must have been stable and may not have had 2 or more of the following laboratory parameters associated with decompensated liver disease: conjugated bilirubin > 1.5 x the upper limit of the normal range (ULN), prothrombin time > 1.5 x ULN, platelets < 60,000/mm^3, serum albumin < 3.0 g/dL
* Must have had at least 12 weeks of center-specific prophylactic therapy including hepatitis B immunoglobulin (HBIg) posttransplant
* Calculated creatinine clearance ≥ 40 mL/min using the Cockcroft-Gault equation
* No significant evidence of ongoing deterioration of renal function
* Negative serum beta-human chorionic gonadotropin (for females of childbearing potential only)

Exclusion Criteria:

* Subjects with HBV recurrence, ie, confirmed HBV DNA ≥ 400 copies/mL, following liver transplant
* Pregnant women, women who were breast feeding or who believed they may have wished to become pregnant during the course of the study
* Males and females of reproductive potential who were unwilling to use an effective method of contraception during the study and for at least 30 days from the date of last dose of study drug
* Evidence of hepatocellular carcinoma (HCC), eg, alpha-fetoprotein > 50 ng/mL, or by any other standard of care measure or presence of multifocal HCC at the time of transplantation if transplantation was within 144 weeks of screening
* Prior TDF or FTC/TDF experience post-transplant or > 12 months treatment with TDF or FTC/TDF treatment pretransplant
* Coinfection with hepatitis C virus (by serology), HIV, or hepatitis D virus pretransplant or at screening
* Significant renal, cardiovascular, pulmonary, or neurological disease
* Known hypersensitivity to the study drugs, the metabolites, or formulation excipients
* Were likely to receive systemic drugs with nephrotoxic potential, except immunosuppressive agents (eg, cyclosporine, tacrolimus), during the course of the study
* History of variceal bleeding or hepatic encephalopathy following orthotopic liver transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Teperman, MD, Principal Investigator — NYU Langone Health
Locations (5):
- United States (5):
  - Los Angeles, California
  - San Francisco, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 7 sites in the United States. The first participant was screened on 12 September 2007. The last participant observation was on 03 May 2011.
Pre-assignment Details: 51 participants were screened; 40 received emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF)+HBIg in the pre-randomization period; 37 received FTC/TDF+HBIg or FTC/TDF in the randomized period.
Groups:
- FTC/TDF+HBIg: For the Participant Flow, this group includes all participants who received any treatment in the pre-randomization period, and participants who received FTC/TDF+HBIg in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- FTC/TDF: For the Participant Flow, this group includes participants who received FTC/TDF in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily.
Period: Pre-Randomization Period
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Started | 40 | 0
Completed | 37 | 0
Not Completed | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Randomized Period
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Started | 19 (19 of 37 participants who completed the pre-randomization period were randomized to FTC/TDF+HBIg.) | 18 (18 of 37 participants who completed the pre-randomization period were randomized to FTC/TDF.)
Completed | 18 | 16
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Three groups are reported for baseline characteristics: the 2 treatment groups in the randomized period, and non-randomized participants who discontinued prior to the randomized period.
Groups:
- FTC/TDF+HBIg: For Baseline Characteristics, this group includes participants who received FTC/TDF+HBIg in the pre-randomization period, and were then randomized to receive FTC/TDF+HBIg in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- FTC/TDF: For Baseline Characteristics, this group includes participants who received FTC/TDF+HBIg in the pre-randomization period, and were then randomized to receive FTC/TDF in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- Not Randomized: For Baseline Characteristics, this group includes participants who received FTC/TDF+HBIg in the pre-randomization period only. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- Total: Total of all reporting groups
Arm/Group | FTC/TDF+HBIg | FTC/TDF | Not Randomized | Total
Number analyzed (Participants) | 19 | 18 | 3 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9.7) | 59 (9.1) | 64 (6.0) | 57 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 15 | 15 | 2 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 17 | 16 | 3 | 36
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 6 | 8 | 1 | 15
  White | 7 | 5 | 1 | 13
  Black | 5 | 4 | 1 | 10
  Other | 1 | 1 | 0 | 2
Baseline hepatitis B virus (HBV) DNA Below 169 copies/mL [Number; unit: participants]
  < 169 copies/mL | 19 | 18 | 3 | 40
  ≥ 169 copies/mL | 0 | 0 | 0 | 0
Baseline alanine aminotransferase (ALT) above the upper limit of the normal range (ULN) [Number; unit: participants] — The upper limit of the normal range (ULN) for ALT was 34 U/L for females 18-69 years of age, and 32 U/L for females over age 69; the ULN was 43 U/L for males 18-69 years of age, and 35 U/L for males over age 69.
  participants
    > ULN | 0 | 2 | 0 | 2
    ≤ ULN | 19 | 16 | 3 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HBV Recurrence Prior to or at Week 72
Description: HBV recurrence was defined as either HBV DNA ≥ 400 at 2 consecutive visits before Week 72, or HBV DNA ≥ 400 at the Week 72 visit.
Time Frame: Pretreatment baseline through Week 72
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Groups:
- FTC/TDF+HBIg: Participants received FTC/TDF+HBIg for up to 24 weeks in the pre-randomization period; those who completed 24 weeks of treatment were then randomized to receive FTC/TDF+HBIg in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- FTC/TDF: Participants received FTC/TDF+HBIg for up to 24 weeks in the pre-randomization period; those who completed 24 weeks of treatment were then randomized to receive FTC/TDF in the randomized period. FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 19 | 18
percentage of participants | 0 | 0

2. Secondary Outcome: Percentage of Participants With HBV Recurrence at Week 96
Description: HBV recurrence was defined as HBV DNA ≥ 400 at the Week 96 visit.
Time Frame: Week 96
Population: Participants in the Full Analysis Set with available data at Week 96 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 17 | 16
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Subjects With HBV DNA < 169 Copies/mL at Week 72
Time Frame: Week 72
Population: Participants in the Full Analysis Set with available data at Week 72 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 19 | 16
percentage of participants | 100 | 100

4. Secondary Outcome: Percentage of Participants With HBV DNA < 169 Copies/mL at Week 96
Time Frame: Week 96
Population: Participants in the Full Analysis Set with available data at Week 96 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 17 | 16
percentage of participants | 100 | 100

5. Secondary Outcome: Percentage of Participants With Normal ALT at Week 72
Description: Range of normal ALT was 6 to 34 U/L for females 18-69 years of age, and 6 to 32 U/L for females over age 69. Range of normal ALT was 6 to 43 U/L for males 18-69 years of age, and 6 to 35 U/L for males over age 69.
Time Frame: Week 72
Population: Participants in the Full Analysis Set with available data at Week 72 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 19 | 16
percentage of participants | 89 | 81

6. Secondary Outcome: Percentage of Participants With Normal ALT at Week 96
Description: as for outcome 5
Time Frame: Week 96
Population: Participants in the Full Analysis Set with available data at Week 96 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF+HBIg | FTC/TDF
Number analyzed (Participants) | 17 | 15
percentage of participants | 88 | 80

ADVERSE EVENTS:
Time Frame: Pretreatment baseline to Week 96
Description: Adverse events are presented for 3 reporting groups: a single group of all participants who were enrolled and received FTC/TDF+HBIg in the 24-week pre-randomization period, and 2 groups (FTC/TDF with or without HBIg) in the 72-week randomized period that followed.
Groups:
- FTC/TDF+HBIg, Pre-randomization Period: For the reporting of Adverse Events, this group includes participants who received FTC/TDF+HBIg during the pre-randomization period, and were analyzed from pretreatment baseline to Week 24 (pre-randomization period). FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- FTC/TDF+HBIg, Randomized Period: For the reporting of Adverse Events, this group includes participants who received FTC/TDF+HBIg during the randomized period, and were analyzed from randomization (at the Week 24 visit) to Week 96 (randomized period). FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
- FTC/TDF, Randomized Period: For the reporting of Adverse Events, this group includes participants who received FTC/TDF during the randomized period, and were analyzed from randomization (at the Week 24 visit) to Week 96 (randomized period). FTC (200 mg)/TDF (300 mg) was administered as a fixed-dose combination tablet orally once daily. HBIG was administered according to site-specific protocols.
Arm/Group | FTC/TDF+HBIg, Pre-randomization Period | FTC/TDF+HBIg, Randomized Period | FTC/TDF, Randomized Period
Serious Adverse Events (participants affected / at risk) | 2/40 | 6/19 | 3/18
Other Adverse Events (participants affected / at risk) | 22/40 | 15/19 | 11/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/TDF+HBIg, Pre-randomization Period (N=40) | FTC/TDF+HBIg, Randomized Period (N=19) | FTC/TDF, Randomized Period (N=18)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Liver transplant rejection (Immune system disorders) | 0 | 1 | 0
Transplant rejection (Immune system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FTC/TDF+HBIg, Pre-randomization Period (N=40) | FTC/TDF+HBIg, Randomized Period (N=19) | FTC/TDF, Randomized Period (N=18)
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 5 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Creatine renal clearance decreased (Investigations) | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 1
Headache (Nervous system disorders) | 2 | 2 | 1
Pharyngolarylngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0
Bronchiectasis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 3 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Chest pain (General disorders) | 0 | 1 | 0
Noncardiac chest pain (General disorders) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1 | 1
Cardiac murmur (Investigations) | 0 | 1 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0
Seasonal allergies (Immune system disorders) | 0 | 2 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0
Vein disorder (Vascular disorders) | 0 | 1 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Pollakiurua (Renal and urinary disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Adrenal disorder (Endocrine disorders) | 0 | 1 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years